CLINICAL TRIAL: NCT04316845
Title: 18F-Fluorocholine PET/CT in the Pre-operative Localization of Hyperfunctional Parathyroid Gland in Primary and Secondary Hyperparathyroidism
Brief Title: 18F-fluorocholine PET/CT for Hyperparathyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB106-74-A
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2020-03

CONDITIONS: Hyperparathyroidism
Keywords: Hyperparathyroidism; sestamibi; scintigraphy; 18F-Fluorocholine, PET
MeSH Terms: conditions — Hyperparathyroidism

STUDY DESIGN:
Intervention Model Description: Patient undergoes both 18F-fluorocholine PET/CT and sestamibi scan
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-fluorocholine PET/CT (Experimental): 18F-fluorocholine PET/CT
  Interventions: Diagnostic Test: 18F-fluorocholine PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-fluorocholine PET/CT — Patients undergo both 18F-fluorocholine PET/CT and Single isotope dual phase Tc-99m sestamibi scan (both planar scan and SPECT/CT)
  Other Names: Tc-99m sestamibi scintigraphy

SUMMARY:
Hyperparathyroidism is a common endocrine disorder which can result in many severe complications. For patients with hyperparathyroidism, Tc-99m sestamibi imaging is the major imaging tool for pre-operative localization of the hyperfunctioning gland. However, sestamibi scan have only limited sensitivity in detecting multigland disease and hyperplastic foci. New imaging tracer with 18F-fluorocholine (18F-FCH) has showed avidity in parathyroid tissues. Nevertheless, the research data of 18F-FCH PET/CT are only preliminary.

The goal of our study is to compare the diagnostic performance of 18F-FCH PET/CT and single isotope dual phase sestamibi scintigraphy for patients with hyperparathyroidism.

From Jan. 1st, 2018 till Dec. 31st, 2019, the investigators will prospectively enroll patients with biochemical evidence of hyperparathyroidism and intended to receive pre-operative image study. The patients will receive single isotope dual phase sestamibi scintigraphy and 18F-FCH PET/CT. Each image will be evaluated by experienced interpreter for abnormal uptake suspicious for hyperfunctioning parathyroid gland. The reference standard will be the final surgical results. Diagnostic performance of both sestamibi scan and PET/CT scan will be measured and calculated.

DETAILED DESCRIPTION:
The investigators conducted a prospective study to investigate the performance of 18F-choline (FCH) PET/CT and 99mTc- sestamibi scintigraphy in the pre-operative localization of hyperfunctioning parathyroid glands.

Single isotope dual phase Tc-99m sestamibi imaging protocol:

Fasting is not needed before radiotracer injection. No specific drug restriction is needed. Scan will be conduced by using a dual head gamma camera unit (Infinia Hawkeye; GE Medical Systems, Milwaukee,Wis), and scans will be interpreted on a work station with the use of compatible software (Xeleris).

An indwelling intravenous catheter connected to an infusion line and an saline syringe will be set on each patient. 99mTc-sestamibi (925 +/- 10% MBq) will be injected intravenously through the infusion line and will be flushed by saline. The image acquisition of the first phase is to be taken 15 minutes after radiotracer injection. The second phase will be acquired 2-4 hours after the initial tracer injection. The scintigraphic scan field will cover from neck to chest. Additional field-of-view will be performed if the patient has known surgically reimplanted parathyroid gland in the arms.

Two nuclear medicine physicians assess the single isotope dual phase 99mTc-sestamibi scintigraphy. The investigators have access to the patients' history and interpreted individually by each reader, with disagreements to be resolved by consensus. Uptake conspicuity will be evaluated in 4-graded scale. 0. Unable to identify any focal uptake; 1. Inconspicuous focus; 2. Focal mild uptake; 3. Focal intense uptake. For the determination of a diagnosis, score 0 and 1 are considered a negative resulte and 2 to 3 a positive result.

18F-FCH PET imaging protocol: Fasting is not needed before radiotracer injection. No specific drug restriction is needed. Scan will be conduced by using a PET/CT unit (Discovery ST; GE Medical Systems, Milwaukee,Wis), and scans will be interpreted on a work station with the use of compatible software (Xeleris).

An indwelling intravenous catheter connected to an infusion line and an saline syringe will be set on each patient. 18F-FCH (185 +/- 10% MBq) will be injected intravenously through the infusion line and will be flushed by saline. The injected 18F-FCH dose, injection time, post-injection residual activity, time of start imaging and time of end imaging will be recorded on case report form. 18F-FCH PET/CT scan acquisition is to be taken 5 to 10 minutes after radiotracer injection. The PET/CT (80-120 mA, 120 kVp) scan field will cover from skull to mid-thigh. Patient with reimplanted focus will be put into the field-of-view. The 18F-FCH PET/CT scan time will require 35-40 minutes.

Two nuclear medicine physicians assess the 18F-FCH PET/CT images. The investigators have access to the patients' history and interpreted individually by each reader, with disagreements to be resolved by consensus. However, the interpreters have no access to the sestamibi imaging results. For 18F-FCH PET/CT images, uptake conspicuity will be evaluated in 4-graded scale. 0. Unable to identify any focal uptake; 1. Inconspicuous focus; 2. Focal mild uptake; 3. Focal intense uptake. For the determination of a diagnosis, score 0 and 1 are considered a negative resulte and 2 to 3 a positive result.

Reference standard is established by surgical pathology:

The reference standard will be the surgical pathological results. Removed gland will be histologically confirmed as parathyroid adenoma or hyperplasia. For in situ hyperfunctioning parathyroid glands, the image results will be compared with the surgical results as correct lateralization (right side or left side), and correct polarity (upper pole or lower pole), sequentially. For ectopic and reimplanted glands, presence of pathological or biochemical evidence of hyperfunctioning gland removal of the image suggested lesion will be the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are diagnosed to have hyperparathyroidism based on serum iPTH data (> 72 pg/mL).
2. Planned to undergo surgical resection of the hyperfunctioning parathyroid gland.
3. Referred for single isotope dual phase Tc-99m sestamibi scintigraphy.
4. The 18F-FCH PET is performed within 6 weeks of the single isotope dual phase Tc-99m sestamibi scintigraphy.
5. If premenopausal and sexually active woman, need contraception (tubal ligation, intrauterine devices, or oral contracepts/condom after the last menstrual period till the image exams)

Exclusion Criteria:

1. Surgical management is not considered.
2. Younger than 20-year-old.
3. Factors that hampers the patient to receive positron emission tomography, e.g., unstable vital signs (shock), conscious disturbance, claustrophobia, etc...
4. Allergic to investigaional drug.
5. Pregnant or lactating woman.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The sensitivities of 18F-fluorocholine PET/CT and 99mTc sestamibi scan | 6 weeks
  The lesion-based sensitivities of these two image modalities using surgical pathology of the parathyroid gland as reference standard (The number of true positive image findings/The number of pathologically confirmed parathyroid adenoma or hyperplasia)
The specificities of 18F-fluorocholine PET/CT and 99mTc sestamibi scan | 6 weeks
  The lesion-based specificities of these two image modalities using surgical pathology of the parathyroid gland as reference standard (The number of true negative image findings/The number of negative finding on surgical pathology)
The accuracies of 18F-fluorocholine PET/CT and 99mTc sestamibi scan | 6 weeks
  The lesion-based accuracies of these two image modalities using surgical pathology of the parathyroid gland as reference standard (True positive and true negative image findings/The number of all surgical specimens)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hsin Liu, M.D., Principal Investigator — Hualien Tzu Chi Hospital, Buddhist Tzu ChiMedical Foundation
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen YH, Chen HT, Lee MC, Liu SH, Wang LY, Lue KH, Chan SC. Preoperative F-18 fluorocholine PET/CT for the detection of hyperfunctioning parathyroid glands in patients with secondary or tertiary hyperparathyroidism: comparison with Tc-99m sestamibi scan and neck ultrasound. Ann Nucl Med. 2020 Aug;34(8):527-537. doi: 10.1007/s12149-020-01479-2. Epub 2020 May 20. PMID 32436180